CLINICAL TRIAL: NCT06116721
Title: Evaluation of the Frequency of APOL1 Gene Variants in Kidney Donors and the Impact of These Variants on the Long-term Renal Function of Kidney Transplant Donors and Recipients
Brief Title: Evaluation of APOL1 Gene Variants in Kidney Donors and Their Impact on Long-term Renal Function in Donors and Recipients
Status: Recruiting | Type: Observational
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Helio Tedesco Silva Junior, Principal Investigator, Hospital do Rim e Hipertensão
Other Study IDs: Hospital do Rim - FOR
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Kidney Diseases; Transplant Failure
Keywords: APOL1 gene; Kidney transplantation; Living donor; Kidney function; Kidney graft survival
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — High-risk variants of the APOL1 gene: they are homozygous (G1 / G1 or G2 / G2) and compound heterozygous (G1 / G2) forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the frequency of APOL1 gene variants in kidney donors and the impact of these variants on the long-term renal function of kidney transplant donors and recipients.

DETAILED DESCRIPTION:
Introduction: Chronic kidney disease (CKD) is a worldwide public health problem and kidney transplantation, when indicated, is the treatment of choice for CKD. Kidney transplant survival at the end of the first year is greater than 95%, however, there has not been a corresponding improvement in long-term kidney graft survival outcomes. Factors such as acute or chronic rejection, bacterial or viral infections, de novo or recurrent glomerulopathies are associated with worsening kidney function in the long term. Genetic variants of the Apolipoprotein L1 (APOL1) gene present in individuals with African ancestry (AF) may also interfere with transplant results. In the general population, individuals with SCA have a higher risk of CKD and one of the most accepted hypotheses is that the APOL1 gene is associated with CKD. Genetic variants (G1 and G2) are exclusive to individuals with SCA and confer a higher risk of CKD. In the transplant population, kidneys from deceased donors of African ancestry (AF) with genetic variants of the APOL1 gene have worse renal graft survival. Recipients with the genetic variants, regardless of donor genotype, are at increased risk of rejection and graft loss by immune-mediated mechanisms that damage the kidney through activation of T and NK cells. In Brazil, more than 5000 transplants are performed per year and it is one of the countries outside Africa with the highest number of Afro-descendants, a high rate of miscegenation and a high prevalence of African ancestry. Despite this, there are no studies on the frequency of APOL1 gene variants in this population, as well as their impact on the clinical evolution of kidney transplantation. General objective: To evaluate the association between APOL1 gene risk variants and long-term renal function in living donors and their respective recipients. Specific objectives: i - To measure the prevalence of APOL1 gene variants in the population of living kidney donors; ii - Evaluate the impact of the presence of APOL1 gene risk variants in living kidney donors, on renal graft survival in their respective recipients; iii- To verify the impact of the presence of risk variants of the APOL1 gene on the long-term renal function of living kidney donors after nephrectomy for donation. Methodology: Evaluation of recipients: longitudinal, observational, retrospective cohort study. Adult kidney transplant recipients from a living donor will be included, who have undergone the transplant at the Hospital do Rim in the period between January 1, 2008 and March 31, 2015, and who remained alive and with a functioning graft one year after the transplant. . The observation period will be until March 2020 (five years). The following will be excluded: recipients who have previously undergone transplantation of other organs and recipients who were transferred for follow-up in other centers before 12 months of follow-up after the transplant was performed. Donor evaluation: cross-sectional cohort study in donors who donated a kidney in the period between January 1, 2008 and March 31, 2015. The prevalence of APOL1 gene variants in this population will be determined and clinical information will be evaluated of the donors, from the date of the nephrectomy until the moment of collection of the exams. In the period covered, 2152 transplants were performed with a living donor. It is estimated that the prevalence of APOL1 gene variants is between 8 and 13%, including populations with chronic kidney disease and who underwent kidney transplantation. To calculate the sample number, it will be assumed, by hypothesis, to find a difference of 10 ml/min/1.73m2 in the mean Estimated Glomerular Filtration Rate (eGFR) at the end of 5 years between recipients of kidneys from donors who present some risk mutation (recessive model) compared with those who do not have any risk mutation. To prove this average in the eGFR, the minimum number required is 98 individuals in each group. It will be assumed that the minimum frequency of mutations is 8% in the population of interest, to reach 98 individuals in each group, the total number of individuals required to be evaluated for the presence of mutation will be 1225 donors. Considering that there will be a loss of follow-up of 20% of the total number of individuals, the total number of donors required to be invited will be 1,535 patients. By including 1,225 donors, 1,225 recipients will be included, totaling 2,450 individuals. Primary endpoint: eGFR 5 years after transplantation in recipients. Secondary endpoints: eGFR decay rate between 1 and 5 years after kidney transplantation in recipients; Graft loss in up to 5 years of follow-up; Death in recipients within 5 years of follow-up; Acute rejection. Exploratory outcomes: current eGFR in donors.

ELIGIBILITY:
Inclusion Criteria:

1.1.1.1. Inclusion criteria 1.1.1.2. For recipients:

1. Living donor kidney transplant recipients, performed at Hospital do Rim from January 1, 2008 to March 31, 2015;
2. Recipients Who have reached one year after the transplant, with a functioning renal graft;
3. Recipients whose donors were located agreed to participate in the research, signed the informed consent form (TCLE) and submitted to the collection of exams.

For donors:

1. Living kidney donors whose donation was made at the Hospital do Rim in the period between January 2008 and December 2015;
2. That they are alive at the time the study begins;
3. Who have signed the TCLE.

Exclusion Criteria:

* For recipients:

  1. Recipients who have undergone the transplant under the age of 18 years;
  2. Recipients who have previously undergone transplantation of other organs; 1.1.3.3. For donors: Donors Who withdraw the informed consent form at any stage of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1.1.2.For evaluation of living donor kidney transplant recipients It will be a longitudinal, observational, retrospective cohort study. Adult kidney transplant recipients from a living donor will be included, who have performed the transplant at the Hospital do Rim in the period between January 1, 2008 and March 31, 2015, who remained alive and with a functioning graft one year after the transplant. The observation time will be until March 2020, so that all recipients have had the opportunity to complete at least 5 years of follow-up after transplantation.
Sampling Method: Probability Sample
Enrollment: 2450 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
For evaluation of living donor kidney transplant recipients | 12 months
  It will be a longitudinal, observational, retrospective cohort study. Adult kidney transplant recipients from a living donor will be included, who have performed the transplant at the Hospital do Rim in the period between January 1, 2008 and March 31, 2015, who remained alive and with a functioning graft one year after the transplant. The observation time will be until March 2020, so that all recipients have had the opportunity to complete at least 5 years of follow-up after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gaspar Tavares, Study Director — Medical Physician; Helio Tedesco Silva Junior, Principal Investigator — Doctor of Renal Transplant Unit; Mônica Rika Nakamura, Study Chair — Study coordinator
Locations (1):
- Hospital do Rim, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No